CLINICAL TRIAL: NCT03955900
Title: Latin American Multiple Myeloma Registry Study
Brief Title: A Registry Study of Participants With Multiple Myeloma in Latin America
Acronym: MYLACRE
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108622; 54767414MMY4021 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2019-05-17; First posted 2019-05-20 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Multiple Myeloma (MM): Participants with MM will be observed in real-world clinical practice settings. The primary data source for this study will be the medical records of each participant.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Both retrospective and prospective data will be collected. The retrospective data will be collected through medical chart review.

SUMMARY:
The purpose of this study is to characterize the multiple myeloma (MM) population concerning demographics and clinical characteristics (for example. frailty, risk strata, manifestations of target organ damage [TOD]) in 6 countries (that is Argentina, Brazil, Mexico, Chile, Colombia and Panama); and to profile the treatment landscape of Latin American MM participants, including factors associated with health-care provider (HCP) selections of different treatment regimens. These factors can include a participant's demographic and clinical characteristics and availability of different therapy options per institution in each country.

ELIGIBILITY:
Inclusion Criteria:

* Incident diagnosis of MM between 01 January 2016 and 31 December 2020 (that is the first observed diagnosis noted in the medical charts)
* An informed-consent form (ICF) or participation agreement must be signed before any data are collected only if a waiver is not permissible. For deceased participants who did not provide consent before death, the permission to research on their information should satisfy the local requirements (that each study site's ethics committee and each country's regulatory authority)

Exclusion Criteria:

* Failed to satisfy one or more of the foregoing inclusion criteria or
* Only with diagnosis of smouldering myeloma between 01 January 2016 and 31 December 2020 in the medical charts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Multiple Myeloma (MM)
Sampling Method: Probability Sample
Enrollment: 2059 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Demographic Characteristics of Multiple Myeloma (MM) Participants | Baseline
  Demographic characteristics (such as age, gender, race, ethnicity, country of residence, and health insurance) of MM participants will be assessed at baseline.
Number of Participants with Comorbid Conditions | Baseline
  Number of participants with comorbid conditions (such as obesity, diabetes, cardiovascular disease, anemia alcohol, and tobacco use) will be assessed at baseline.
General Health Status Based on Frailty Score | Approximately up to 2.7 years
  General health status based on Frailty Score will be reported. International Myeloma Working Group (IMWG) frailty score: Participants frailty status will be assessed on the basis of 4 components: age (less than [<75], 76- 80, and greater than [>]80 years correspond to frailty scores of 0, 1, and 2, respectively), the charlson comorbidity scoring system without age weighting (scores of less than or equal to [<=]1 and greater than or equal to [>=]2 correspond to frailty scores of 0 and 1, respectively), independence in activities of daily living (scores of >4 and <=4 correspond to frailty scores of 0 and 1, respectively) and instrumental activities of daily living scale (scores of >5 and <=5 correspond to frailty scores of 0 and 1, respectively). The sum of the 4 frailty scores equals the total frailty score. The total frailty score ranges from 0 to 5, with a total of three categories: 0 (fit), 1 (intermediate-fitness) and greater than or equal to (>=)2 (frail).
Eastern Cooperative Oncology Group (ECOG) Performance Status Score | Approximately up to 2.7 years
  ECOG performance status is a standard criterion for measuring how the disease impacts daily living abilities. It describes the level of functioning in terms of the ability to care for oneself, daily activity, and physical ability (walking, working, etc). ECOG performance status score ranges from Grade 0 to 5: 0= Fully active and performances without restriction, 1= Restricted in physically strenuous activity, 2= Ambulatory and capable of all self-care but unable to carry out any work activities, 3= Capable of only limited self-care and confined to bed or chair more than 50% of waking hours, 4= Completely disabled, and 5= Dead.
Sequence of Treatments in Participants with Multiple Myeloma (MM) | Approximately up to 2.7 years
  Treatment sequences for participants with MM within routine clinical care will be assessed.
Number of Participants in Each Stage of Multiple Myeloma (MM) Disease | Approximately up to 2.7 years
  Number of participants in each stage of MM disease will reported. The stage of MM disease will be determined by International Staging System (ISS). ISS categorizes MM participants into three groups (Stage I, II, or III). Stage I: beta2-microglobulin less than (<)3.5 milligram per liter (mg/L) and albumin greater than or equal to (>=)3.5 gram (g)/100 milliliter (mL); stage II: neither stage I nor stage III; and stage III: beta2-microglobulin >=5.5 mg/L.

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately up to 2.7 years
  The OS in MM participants will be measured and reported from diagnosis to the date of death.
Progression-Free Survival (PFS) | Approximately up to 2.7 years
  PFS is defined as time from diagnosis to disease progression. IMWG criteria for disease progression: increase of greater than or equal to (>=)25 percent (%) from lowest response value in any one of the following: Serum M-component (absolute increase must be >=0.5 gram per deciliter [g/dL]), Urine M-component (absolute increase must be >=200 milligram per 24 hour [mg/24 hour]), only in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain levels (absolute increase must be greater than >10 mg/dL), Bone marrow plasma cell percentage: the absolute percent must be >=10%, Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas, Development of hypercalcemia (corrected serum calcium >11.5 mg/dL or 2.65 millimoles per liter [mmol/L]) that can be attributed solely to the plasma cell proliferative disorder.
Percentage of Participants with Complete Response (CR) | Approximately up to 2.7 years
  Complete response (CR) per International Myeloma Working Group (IMWG 2014) criteria is defined by negative immunofixation on the serum and urine, disappearance of any soft-tissue plasmacytomas, and less than (<)5 percent (%) plasma cells in bone marrow.
Percentage of Participants with Stringent Complete Response (sCR) | Approximately up to 2.7 years
  Stringent CR per IMWG criteria is defined by a below plus normal fee-light-chain (FLC) ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence.
Duration of Response | Approximately up to 2.7 years
  Duration of response is defined as the time from the date of initial documentation of a response (CR or partial response [PR]) to the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death. Relapse as per IMWG criteria is defined as presence of definite new bone lesions and/or soft-tissue plasmacytomas, with a clear increase in the size of existing plasmacytomas, or hypocalcemia that cannot be attributed to another cause.
Time to Next Treatment | Approximately up to 2.7 years
  Time to next treatment is defined as the time from diagnosis to the start of the next-line treatment.
Percentage of Participants who Adopted Treatment Regimens | Approximately up to 2.7 years
  Percentage of participants who adopted treatment regimens will be reported.
Number of Participants with Adverse Events | Approximately up to 2.7 years
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants who Underwent Different Types of Minimal Residual Disease (MRD) Tests | Approximately up to 2.7 years
  Number of participants who underwent different types of MRD tests will be reported. MRD tests include next-generation [NG] flow cytometry, NG sequencing, positron emission tomography with computed tomography [PET-CT].

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (22):
- Argentina (5):
  - Fundaleu, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Instituto de Oncologia Angel H. Roffo, Buenos Aires
  - Hospital Privado - Centro Medico de Cordoba, Córdoba
  - Hospital Italiano de La Plata, La Plata
- Brazil (9):
  - Fundacao para o Desenvolvimento Medico Hospitalar (UNESP Botucatu), Botucatu
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - CEHON, Salvador
  - Clinica Sao Germano, São Paulo
  - Fundação Antônio Prudente - A.C. Camargo Cancer Center, São Paulo
  - SPDM - Associacao Paulista para o Desenvolvimento da Medicina - Hospital Sao Paulo, São Paulo
  - Instituto de Assistencia Medica ao Servidor Publico Estadual - IAMSPE, São Paulo
- Colombia (5):
  - Hospital Universitario Mayor - Mederi, Bogotá
  - Fundacion Santa Fe de Bogota, Bogotá
  - Clinica de Occidente, Cali
  - Fundacion Oftalmologica de Santander - FOSCAL, Floridablanca
  - Hospital Pablo Tobon Uribe, Medellín
- Mexico (2):
  - Centro de Investigación Farmacéutica Especializada, Guadalajara
  - Hospital Angeles Lomas, Huixquilucan
- Centro Hemato Oncologico Paitilla, Panama City, Panama

REFERENCES:
- [Derived] Hungria V, Gaiolla R, Galvez K, Remaggi G, Schutz N, Bittencourt R, Maiolino A, Quintero-Vega G, Cugliari MS, Braga WMT, Villarim CC, Crusoe E, Enrico AI, Caiero G, Bigonha J, Moura FL, Figueroa J, Sossa Melo CL, Lombana M, Pei H, Fernandez M, Saes J, Trufelli DC. Health care systems as determinants of outcomes in multiple myeloma: final results from the Latin American MYLACRE study. Blood Adv. 2025 Mar 25;9(6):1293-1302. doi: 10.1182/bloodadvances.2024013838. PMID 39657126